CLINICAL TRIAL: NCT02327741
Title: Evaluation of Safety, Benefits and Complications of Long-term Dual Antiplatelet Therapy in Patients With Angioplasty
Brief Title: Efficacy of Long Term Plavix Therapy Post Angioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 90-2348
Record Dates: First submitted 2014-12-13; First posted 2014-12-30 (Estimated); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Dual antiplatelet therapy; clopidogrel; percutaneous coronary intervention
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- plavix long term (Experimental): taking plavix more than 12 months
  Interventions: Drug: plavix
- plavix short term (Active Comparator): taking plavix less than 12 months
  Interventions: Drug: plavix

INTERVENTIONS:
Drug: plavix — taking plavix more than 12 months
  Arms: plavix long term
Drug: plavix — taking plavix less than 12 months
  Arms: plavix short term

SUMMARY:
1010 patients post stenting were enrolled to receive Plavix more than 12 months and less than that and rate of bleeding, complication and major cardiovascular adverse events ( MACE) were compared to evaluate safety and feasibility of long term Plavix therapy post stenting.

DETAILED DESCRIPTION:
1010 patients from registry of angioplasty and stenting in Shiraz and Baghiatolah hospital were enrolled and long term Plavix therapy more than and less than 12 months were compared between two groups of patients prospectively and rate of major adverse cardiovascular events ( MACE) (death, myocardial infarction, cerebrovascular accidents and revascularization) and rate of bleeding were compared between 2 groups.Syntax score and American heart association ( AHA) score of coronary involvement were measured and MACE was compared to these scores.

ELIGIBILITY:
Inclusion Criteria:

* post stent ( lesion more than 70% and vessel more than 2.25 mm )

Exclusion Criteria:

* allergy to acetylsalicylic acid or clopidogrel,
* planned surgery within 24 months of percutaneous coronary intervention unless the dual antiplatelet therapy could be maintained throughout the perisurgical period
* history of bleeding diathesis
* major surgery within 15 days
* active bleeding
* previous stroke in the past 6 months
* concomitant or foreseeable need for oral anticoagulation therapy
* pregnancy, life expectancy <24 months, participation in another trial
* inability to provide informed consent

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: javad kojuri, M.D. M.S., Principal Investigator — shiraz university of medcal sciences

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plavix Short Term | Plavix Long Term
Started | 502 | 508
Completed | 502 | 508
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plavix Long Term | Plavix Short Term | Total
Number analyzed (Participants) | 508 | 502 | 1010
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10) | 60.1 (10) | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 180 | 364
  Male | 324 | 322 | 646
type of stents [Count of Participants; unit: Participants]
  drug eluting stents | 328 | 327 | 655
  metallic stents | 180 | 175 | 355
coronary risk factors [Count of Participants; unit: Participants] | 356 | 351 | 707
which coronary vessel involved [Count of Participants; unit: Participants]
  LAD( left anterior descending) | 392 | 400 | 792
  LCX ( left circumflex) | 78 | 80 | 158
  RCA ( right coronary artery) | 38 | 22 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Major Bleeding Need Transfusion
Description: number of patients with major bleeding need transfusion
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Plavix Short Term | Plavix Long Term
Number analyzed (Participants) | 502 | 508
Participants | 7 | 10

2. Primary Outcome: Number of Patients With Myocardial Infarction Need Hospital Admission
Description: The number of patients with myocardial infarction need hospital admission
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Plavix Short Term | Plavix Long Term
Number analyzed (Participants) | 502 | 508
Participants | 5 | 7

3. Primary Outcome: Number of Patients With Central Vascular Accidents Proved by CT Scan
Description: the number of patients with major vascular brain accidents ( CVA) proved by CT scan
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Plavix Short Term | Plavix Long Term
Number analyzed (Participants) | 502 | 508
Participants | 0 | 1

4. Primary Outcome: Number of Patients With Death Due to Cardiac Causes
Description: the number patients with death due to cardiac causes
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Plavix Short Term | Plavix Long Term
Number analyzed (Participants) | 502 | 508
Participants | 0 | 0

5. Primary Outcome: Revascularization - Need for Redo Bypass Surgery and Redo Angioplasty
Description: need for redo bypass surgery and redo angioplasty
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Plavix Short Term | Plavix Long Term
Number analyzed (Participants) | 502 | 508
Participants | 15 | 14

6. Primary Outcome: Number of Patients With Minor Bleeding
Description: the number of patients with petechiae and superficial ecchymosis or nose bleeding need no admission or drug changes
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Plavix Short Term | Plavix Long Term
Number analyzed (Participants) | 502 | 508
Participants | 13 | 4

7. Secondary Outcome: Tolerability - the Number of Patients , Who Are Able to Take Plavix Concerning Compliance and Economic Issues
Description: the number of patients who are able to take plavix concerning compliance and economic issues
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Plavix Short Term | Plavix Long Term
Number analyzed (Participants) | 502 | 508
Participants | 500 | 506

ADVERSE EVENTS:
Arm/Group | Plavix Short Term | Plavix Long Term
All-Cause Mortality (participants affected / at risk) | 1/502 | 1/508
Serious Adverse Events (participants affected / at risk) | 20/502 | 14/508
Other Adverse Events (participants affected / at risk) | 13/502 | 4/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plavix Short Term (N=502) | Plavix Long Term (N=508)
bleeding (Blood and lymphatic system disorders) | 20 (20) | 14 (14)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plavix Short Term (N=502) | Plavix Long Term (N=508)
minor bleeding (Blood and lymphatic system disorders) | 13 (13) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No